CLINICAL TRIAL: NCT01776567
Title: Apposition Assessed Using Optical Coherence Tomography of Chromium Stents Eluting Everolimus From Cobalt Versus Platinum Alloy Platforms.
Acronym: APPOSE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northern Hospital, Australia (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, A/Prof. Peter Barlis, Interventional Cardiologist, Northern Hospital, Australia
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 01/12
Record Dates: First submitted 2012-08-11; First posted 2013-01-28 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; stents; optical imaging
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cobalt Chromium Everolimus-eluting stent (Xience Prime) (Active Comparator): Cobalt Chromium Everolimus-eluting stent (Xience Prime)
  Interventions: Device: Everolimus eluting stents
- Platinum Chromium Everolimus-eluting stent (Promus Element) (Active Comparator): Platinum Chromium Everolimus-eluting stent (Promus Element)
  Interventions: Device: Everolimus eluting stents

INTERVENTIONS:
Device: Everolimus eluting stents

SUMMARY:
The purpose of the trial is to directly compare the Cobalt Chromium platform everolimus-eluting stent, Xience Prime™, with the Platinum Chromium platform everolimus-eluting stent, Promus Element™, in relation to stent scaffolding shape, position with the heart blood vessel and extent of tissue coverage (at 6 months) using optical coherence tomography.

Hypotheses:

1. The alloy composition and strut design of a drug-eluting stent has a direct bearing on stent apposition measured using OCT.
2. Stent design and alloy composition have a direct influence on radial support and scaffold shrinkage.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Symptomatic coronary artery disease including patients with chronic stable angina, silent ischemia, and acute coronary syndromes including non-ST elevation myocardial infarction
3. Presence of one or more coronary artery stenosis > 50% in a native coronary artery with a reference diameter ranging from 2.25 to 4.25 mm which can be covered with one or multiple stents
4. No limitation to the number of treated lesions or number of vessels according to the randomization group
5. De-novo native coronary disease with complex lesions involving: Bifurcations, chronic occlusions > 3 months, lesions > 20mm in length or moderately/heavily calcified lesions of any length

Exclusion Criteria:

1. Known intolerance to aspirin, clopidogrel, heparin, cobalt chromium, platinum chromium, everolimus, contrast material
2. Acute ST-segment elevation myocardial infarction
3. Type A lesion including vessel angulation <45 degrees
4. Bypass graft
5. Inability to provide informed consent
6. Pregnancy
7. Planned surgery within 12 months of PCI unless dual antiplatelet therapy is maintained throughout the peri-surgical period
8. Left ventricular ejection fraction < 25%
9. Serum creatinine > 180mmol/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-12 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
• Percent incomplete stent apposition using OCT of the CoCr-EES versus the PtCr-EES stent inflated to nominal pressure and following optimal post-dilatation. Stent length (mm) at implantation following nominal pressure and following post-dilatation | Immediately following stent deployment

SECONDARY OUTCOMES:
Percentage of uncovered stent struts | 6 mths post initial PCI procedure
Mean neointimal tissue thickness (microns) | 6 months post initial PCI Procedure
Stent length (mm) measured using OCT | 6 months post initial PCI procedure

CONTACTS AND LOCATIONS:
Overall Officials: Peter Barlis, Principal Investigator — Northern Hospital
Locations (4):
- Australia (4):
  - Concord Repatriation Hospital, Concord, New South Wales
  - The Prince Charles Hospital, Brisbane, Queensland
  - Northern Hospital, Epping, Victoria
  - St Vincent's Hospital, Melbourne, Victoria